CLINICAL TRIAL: NCT00181857
Title: Risk of Attention Deficit Hyperactivity Disorder in the Children of Adults With Attention Deficit Hyperactivity Disorder Not Otherwise Specified: A Pilot Study
Brief Title: Risk of Attention Deficit Hyperactivity Disorder (ADHD) in the Children of Adults With ADHD Not Otherwise Specified (NOS)
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Craig B. Surman, MD, Scientific Director of the Adult ADHD Program, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Other Study IDs: 2004-P-002687
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: ADHD
Keywords: ADHD NOS; familial risk; children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Children of Adults with ADHD NOS

SUMMARY:
The researchers plan to explore the validity of the category of ADHD NOS by identifying the risk for ADHD in the children of ADHD NOS adult probands and identifying common correlates of ADHD in these children. The researchers hypothesize that the rate of ADHD will be higher in the children of the ADHD NOS probands than the rate of ADHD previously published for siblings of proband children with ADHD; and ADHD children of ADHD NOS adults will have higher rates of school failure (as measured by their rate of repeated grades, need for tutoring, and placement in special classes) than their non-ADHD siblings.

DETAILED DESCRIPTION:
We plan to explore the validity of the category of ADHD NOS by identifying the risk for ADHD in the children of ADHD NOS adult probands and identifying common correlates of ADHD in these children. We hypothesize the rate of ADHD will be higher in the children of the ADHD NOS probands than the rate of ADHD previously published for siblings of proband children with ADHD; and ADHD children of ADHD NOS adults will have higher rates of school failure (as measured by their rate of repeated grades, need for tutoring, and placement in special classes) than their non-ADHD siblings.

The proposed study includes a one-time fifteen minute survey derived from the ADHD module of the Kiddie Schedule for Affective Disorders - Epidemiological Version (KSADS-E) with the proband of an ADHD NOS study regarding his/her children, in order to assess possible ADHD symptoms of that child. We also ask "school questions" regarding certain aspects of a child's educational experience.

ELIGIBILITY:
Inclusion Criteria:

Must be a biological child of an ADHD NOS proband. The proband must meet the following criterion:

1. Age: above 18 years
2. Sex: male or female
3. Intelligence quotient (IQ) above 80
4. Met criteria for the diagnosis of attention deficit hyperactivity disorder not otherwise specified (ADHD NOS), by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), as manifested in clinical evaluation and confirmed by structured interview. This is operationalized by either:

   * having at least 6 out of 9 current DSM-IV items of either inattention or hyperactivity/impulsivity but < 5 items from either list in childhood, or
   * having 5 out of 9 current DSM-IV items of either inattention or hyperactivity/impulsivity, but not having the 6 current symptoms in either category. This second category will be included independent of the presence or absence of ADHD symptoms in childhood.
5. Had a Clinical Global Impression: ADHD score of 4 (moderately ill) or higher illness severity at a clinical evaluation.
6. Has at least one biological offspring

Exclusion Criteria:

1. No adequate informant is available to answer the survey questions.
2. Sensorimotor deficits. (These include deficits that would impede the survey process, e.g. profound deafness, blindness, inadequate command of the English language, or profound disorders of language.)
3. Psychosis, autism, schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Children of Adults with ADHD NOS
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-02; Primary Completion 2006-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
ADHD Diagnosis | at evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Craig Surman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States